CLINICAL TRIAL: NCT01152099
Title: A Randomized, Controlled Clinical Trial About the Contribution of Manual Lymph Drainage in Complex Physical Therapy for Patients With Lymphoedema Secondary to Mastectomy
Brief Title: A Clinical Trial About the Contribution of Manual Lymph Drainage in Complex Physical Therapy for Patients With Lymphoedema Secondary to Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TFCDLM-07
Record Dates: First submitted 2010-06-24; First posted 2010-06-29 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Lymphoedema
Keywords: Postmastectomy
MeSH Terms: conditions — Lymphedema | interventions — Compression Bandages; Manual Lymphatic Drainage

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GroupA (Active Comparator): Ambulatory treatment is performed during one month. Specific exercises and prevention measures are taught. Multilayer bandage is applied daily during the first four weeks.
  The tailor-made sleeve for lymphedema with gauntlet without protection at the edges and with extension to the shoulder is placed from the first four weeks of treatment. The sleeve is used during the whole day and a night interruption is allowed. Later the patient will continue domiciliary treatment realizing specific exercises for 30 minutes twice a day without fatigue carrying the lymphedema sleeve for at least 12 hours.
  If after three months of treatment a good response is not obtained an ambulatory treatment will be introduced again for one month,and this time the treatment corresponding to the group B or experimental will be applied.
  Interventions: Other: Compression Bandaging
- GroupB (Experimental): Ambulatory treatment is carried out during one month. Specific exercises measures of prevention are taught. MLD is carried out followed by a daily multilayer bandage during the first four weeks. The tailor-made sleeve for lymphedema with gauntlet without protection at the edges and with extension to the shoulder is placed from the first four weeks of treatment. The sleeve is used during the whole day and a night interruption is allowed. Later the patient will continue domiciliary treatment realizing specific exercises for 30 minutes twice a day without fatigue carrying the lymphedema sleeve for at least 12 hours.
  If after three months of treatment a good response is not obtained an ambulatory treatment will be introduced again for one month, and this time the treatment corresponding to the group A or Control will be applied.
  Interventions: Other: Manual Lymph Drainage (MLD) and Compression Bandaging

INTERVENTIONS:
Other: Compression Bandaging — Group A or Control Group: ambulatory treatment is performed during one month. Specific exercises and prevention measures are taught. The tailor-made sleeve for lymphedema with gauntlet without protection at the edges and with extension to the shoulder is placed from the first four weeks of treatment. The sleeve is used during the whole day and a night interruption is allowed. Later the patient will continue domiciliary treatment realizing specific exercises for 30 minutes twice a day without fatigue carrying the lymphedema sleeve for at least 12 hours.
  If after three months of treatment a good response is not obtained an ambulatory treatment will be introduced again for one month,and this time the treatment corresponding to the group B or experimental will be applied.
  Arms: GroupA
Other: Manual Lymph Drainage (MLD) and Compression Bandaging — Specific exercises measures of prevention are taught. MLD is carried out followed by a daily multilayer bandage during the first four weeks. The tailor-made sleeve for lymphedema with gauntlet without protection at the edges and with extension to the shoulder is placed from the first four weeks of treatment. The sleeve is used during the whole day and a night interruption is allowed. Later the patient will continue domiciliary treatment realizing specific exercises for 30 minutes twice a day without fatigue carrying the lymphedema sleeve for at least 12 hours.
  If after three months of treatment a good response is not obtained an ambulatory treatment will be introduced again for one month, and this time the treatment corresponding to the group A or Control will be applied.
  Arms: GroupB

SUMMARY:
Hypothesis:

To know the utility of manual lymph drainage (MLD) as part of the Physical Complex Therapy has turn out relevant because of the exclusive dedication that it supposes to the therapist. To date, the evidence-base for MLD is very limited and only two studies analyze its relevance. The first study measured the effect of compression bandage with or without MLD. The group receiving compression and MLD had a significant reduction in limb volume and decreased pain, despite the fact the MLD was given only for one week (Johansson et al., 1999). A further study investigated the effect of eight sessions of MLD over two weeks in 42 women with breast cancer-related lymphoedema, and the findings suggested that MLD do not contribute significantly to oedema reduction, although the MLD course was relatively short and the study group was limited to those with mild to moderate swelling (20-30 % of difference). Information about the quality of life, using the questionnaire EORT QLQ-C30 was gathered but the results were not considered in the final assessment (Andersen and Cabbage 2000).

Similar studies would provide comparative and enlightening information with regard to the previous results. The investigators could determine if the MLD, in spite of not obtaining an improvement in the volume of the lymphoedema, provides a benefit in the reduction of the symptoms related to it.

The investigators hypothesized that MLD does not contribute significantly in volume limb reduction but it provides a clinical improvement regarding the quality of life according to the questionnaire EORT QLQ-C30.

For the calculation of the sample size the investigators depart from the following assumptions:

The effect of the standard treatment on the control group control will produce an average volume limb reduction of 5 %.

The effect of the treatment in the experimental group will be an average of the 25 % (a minor difference of effects would indicate a discreet effect of the tested treatment). The investigators also assume that, the standard deviation will be similar in both groups and near to 25 %. With this information and for an alpha risk of 0.05 and a power of 0.80 the calculation of the sample size is 20 patients in every group. Considering a rate of withdrawal of 30 % in every group, the appropriate sample size is 58 patients assigned in two groups of 29 patients.

Main aim:

To analyze the effectiveness of Manual Lymph Drainage (MLD) in the treatment of postmastectomy lymphoedema in order to reduce the volume of lymphoedema

Secondary aims:

To analyze the duration of the reduction of the lymphoedema in the time. To analyze the improvement in the concomitant symptomatology of the lymphoedema using the results of two quality of life tests validated in Spanish: EORTC QLQ-C30 version 2.0, for the cancer in general and EORTC QLQ-BR23 specifically for the breast cancer. In particular, the items refering to the upper extremity (47, 48, 49) and to the corporal image (39, 40, 41, 42) and in which the higher the score the worse the result.

Methodology:

Researching Project with methodology of randomized, controlled clinical trial. Group A or Control: patients with standard treatment (care the skin, exercise and measures of compression -bandage for one month and later a sleeve of compression).

Group B or Experimental: patients with standard treatment (care of the skin, exercise and measures of compression (bandage for one month and later a sleeve for lymphoedema) and in addition they receive Manual Lymph Drainage Main variable: Volume reduction of the affected arm after the treatment expressed in percentage.

Number of patients: 58 women.

ELIGIBILITY:
Inclusion Criteria:

* women older than 18 years, intervented of unilateral breast neoplasia with ipsilateral axillar lymphadenectomy
* Patients with ipsilateral lymphoedema with a volume difference of at least 200ml compared to the lateral limb
* Patients who have finished the treatment with Radiotherapy and / or chemotherapy at least six months before the study started
* Informed acceptance has to be signed

Exclusion Criteria:

* Bilateral affectation of both extremities.
* Malignant Active disease
* Acute Lymphoedema (in the first three months postintervention)
* Patients with previous paralysis or vascular alteration in the affected arm
* Patients with a major limitation of 30 º in any of the arches of movement of the ipsilateral shoulder
* Patients with contraindication for Lymphatic Manual Drainage (cellulite, deep venous thrombosis, heart failure, not controlled hypertension, renal failure and important radiodermatitis)
* Patients who have been managed with treatment of rehabilitation in three months previous to the recruitment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2007-09-11 (Actual); Primary Completion 2017-04-24 (Actual); Study Completion 2017-04-24 (Actual)

PRIMARY OUTCOMES:
Statistical analysis | 1 year after the clinical trial ends
  All the patients included in the study will be analyzed and all the analyses will be performed for " intention of treating " except that related to the withdrawal of the treatment that will be done by protocol.
  Firstly an analysis of comparability of the groups using the test of the T de Student or Mann-Withney's Test and test of Fischer´s exact test will be performed. Efficacy analysis:means differences and / or reason of medians for the quantitative variables and reason of risks and NNT for the quantitative variables.

SECONDARY OUTCOMES:
Statistical analysis | 1 year after the clinical trial ends
  Analyses of Safety:side effects and / or withdrawal and / or complications rates.
  In all cases analyses of the confidence intervals will be also calculated.
  Analysis of the Quality of Life

CONTACTS AND LOCATIONS:
Locations (1):
- Rehabilitation Service. Hospital Universitario de La Princesa, Madrid, Spain

REFERENCES:
- [Background] Kopanski Z, Wojewoda T, Wojewoda A, Schlegel-Zawadzka M, Wozniacka R, Suder A, Kosciuk T. Influence of some anthropometric parameters on the risk of development of distal complications after mastectomy carried out because of breast carcinoma. Am J Hum Biol. 2003 May-Jun;15(3):433-9. doi: 10.1002/ajhb.10158. PMID 12704719
- [Background] Johansson K, Lie E, Ekdahl C, Lindfeldt J. A randomized study comparing manual lymph drainage with sequential pneumatic compression for treatment of postoperative arm lymphedema. Lymphology. 1998 Jun;31(2):56-64. PMID 9664269
- [Background] Badger CM, Peacock JL, Mortimer PS. A randomized, controlled, parallel-group clinical trial comparing multilayer bandaging followed by hosiery versus hosiery alone in the treatment of patients with lymphedema of the limb. Cancer. 2000 Jun 15;88(12):2832-7. PMID 10870068
- [Background] Andersen L, Hojris I, Erlandsen M, Andersen J. Treatment of breast-cancer-related lymphedema with or without manual lymphatic drainage--a randomized study. Acta Oncol. 2000;39(3):399-405. doi: 10.1080/028418600750013186. PMID 10987238
- [Background] Harris SR, Hugi MR, Olivotto IA, Levine M; Steering Committee for Clinical Practice Guidelines for the Care and Treatment of Breast Cancer. Clinical practice guidelines for the care and treatment of breast cancer: 11. Lymphedema. CMAJ. 2001 Jan 23;164(2):191-9. PMID 11332311
- [Background] Foldi E, Foldi M, Clodius L. The lymphedema chaos: a lancet. Ann Plast Surg. 1989 Jun;22(6):505-15. doi: 10.1097/00000637-198906000-00007. PMID 2751222
- [Background] Ramos SM, O'Donnell LS, Knight G. Edema volume, not timing, is the key to success in lymphedema treatment. Am J Surg. 1999 Oct;178(4):311-5. doi: 10.1016/s0002-9610(99)00185-3. PMID 10587190
- [Background] McNeely ML, Magee DJ, Lees AW, Bagnall KM, Haykowsky M, Hanson J. The addition of manual lymph drainage to compression therapy for breast cancer related lymphedema: a randomized controlled trial. Breast Cancer Res Treat. 2004 Jul;86(2):95-106. doi: 10.1023/B:BREA.0000032978.67677.9f. PMID 15319562
- [Background] Badger C, Preston N, Seers K, Mortimer P. Physical therapies for reducing and controlling lymphoedema of the limbs. Cochrane Database Syst Rev. 2004 Oct 18;(4):CD003141. doi: 10.1002/14651858.CD003141.pub2. PMID 15495042
- [Derived] Martin ML, Hernandez MA, Avendano C, Rodriguez F, Martinez H. Manual lymphatic drainage therapy in patients with breast cancer related lymphoedema. BMC Cancer. 2011 Mar 9;11:94. doi: 10.1186/1471-2407-11-94. PMID 21392372